CLINICAL TRIAL: NCT06269120
Title: SEMA-CardioDiab HUNGARY: A Multicentre, Prospective, Non-interventional Study to Evaluate Glycemic Control and Weight Changes in Patients With Type 2 Diabetes Initiating Treatment With Oral Semaglutide by Cardiologists or Diabetologists as Part of Local Clinical Practice in Hungary
Brief Title: SEMA-CardioDiab HUNGARY: A Research Study to Understand the Effects of Oral Semaglutide on Blood Sugar Levels, Weight, and Cardiovascular Risk in People With Type 2 Diabetes Patients in Hungary
Status: Recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-7787; U1111-1290-8109 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes: Participants with Type 2 Diabetes (T2D) will initiate oral semaglutide at the discretion of the treating physician, based on approved oral semaglutide label in Hungary and independent from the decision to include the patient in the study.
  Interventions: Drug: Oral Semaglutide

INTERVENTIONS:
Drug: Oral Semaglutide — Patients will be treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician.

SUMMARY:
Participant will get oral semaglutde as prescribed by the study doctor. The study will last for about 26 ± 4 weeks (5 to 7 months). Participant will be asked to complete a questionnaire about how they take oral semaglutide tablets during normal scheduled visit with doctor. Participant will also be asked questions about health and their diabetes treatment and lab tests as part of normal doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/LAR and the treating physician based on local label before and independently from the decision to include the patient in this study.
* Male or female, adults above or equal to 18 years of age at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus.
* Patient on metformin (Met) with or without modern oral antidiabetic (MOAD, that is Dipeptidyl Peptidase-4 Inhibitor [DPP4i] or/and Sodium-glucose cotransporter-2 Inhibitor [SGLT2i]) with or without insulin therapy.
* Available HbA1c value > 7.0% within 90 days prior to the 'Informed Consent and Treatment Initiation visit' (V1) or HbA1c measurement taken in relation with the 'Informed Consent and Treatment Initiation visit' (V1) if in line with local clinical practice.

Exclusion Criteria:

* Previous participation in this study (defined as having given informed consent in this study earlier).
* Treatment with any investigational drug within 30 days prior to enrolment into the study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Glucagon like peptide -1 receptor agonist (GLP1-RA) treatment within 90 days prior to the Treatment Initiation visit (V1).
* Patients diagnosed with type 1 diabetes mellitus.
* Female who is known to be pregnant, undergoing fertility treatment, breastfeeding or intends to become pregnant during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participant diagnosed with T2D and without any prior or current use of oral semaglutide.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c ) reduction greater than or equal to (≥) 0.5%-point and body weight reduction ≥ 5% | From Baseline to end of study (week 32)
  Participants (yes/no).

SECONDARY OUTCOMES:
Change in HbA1c | From Baseline to end of study (week 32)
  Measured in percentage (%)- point.
Change in fasting plasm glucose (FPG) | From Baseline to end of study (week 32)
  Measured in millimoles per liter (mmol/l).
Absolute change in body weight (BW) | From Baseline to end of study (week 32)
  Measured in kilogram (kg).
Relative change in BW | From Baseline to end of study (week 32)
  Measured in %.
HbA1c less than (<) 7.0% | At end of study (week 32)
  Participants (yes/no).
HbA1c <6.5% | At end of study (week 32)
  Participants (yes/no).
Body weight reduction ≥5% | At end of study (week 32)
  Participants (yes/no).
HbA1c reduction ≥1%-point and BW reduction ≥5% | From Baseline to end of study (week 32)
  Participants (yes/no).
HbA1c reduction ≥1%-point and BW reduction ≥3% | From Baseline to end of study (week 32)
  Participants (yes/no).
Change in waist circumference | From Baseline to end of study (week 32)
  Measured in centimeter (cm).
Change in blood pressure (BP) (systolic and diastolic) | From Baseline to end of study (week 32)
  Measured in millimeter of mercury (mmHg).
Change in lipid parameters (total cholesterol, low density lipoprotein cholesterol [LDL-C], high density lipoprotein cholesterol [HDL-C], triglycerides [TG]) | From Baseline to end of study (week 32)
  Measured in mmol/L.
Change in high sensitive C-reactive protein (hsCRP) | From Baseline to end of study (week 32)
  Measured in milligram per liter (mg/l).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Siklósi Kórház, Diabetológia, Siklós, Hungary

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com